CLINICAL TRIAL: NCT06326632
Title: Constant-load Versus Graded Aerobic Exercise for Promoting Cardiorespiratory Fitness and Functional Capacity in Obese Children With Bronchial Asthma: a Randomized Comparative Effectiveness Inquiry
Brief Title: Comparative Effectiveness Study of Constant-Load Versus Graded Aerobic Exercise in Obese Children With Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0022/023
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A prospective, three-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: A single-blind protocol was adopted. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CL-AE group (Experimental): The CL-AE group received a 12-week constant-load aerobic training besides the respiratory retraining program.
  Interventions: Other: Constant-load Aerobic Exercise
- G-AE group (Experimental): The G-AE group received a 12-week intensity- and duration-graded aerobic training in addition to the respiratory re-training.
  Interventions: Other: Graded Aerobic exercise
- Control group (Active Comparator): The control group received the respiratory re-training only for 12 consecutive weeks.
  Interventions: Other: Respiratory Re-training

INTERVENTIONS:
Other: Constant-load Aerobic Exercise — The CL-AE group received a 12-week aerobic training, three times in addition to the respiratory re-training. the program included a moderate-intensity aerobic training program, with an intensity set at 65% of the maximum age-predicted heart rate for 45 minutes. The training intensity and duration were maintained at the same level throughout the program. The CL-AE program included a warm-up for 5 minutes and a cool-down for 5 minutes
  Arms: CL-AE group
Other: Graded Aerobic exercise — The G-AE group received a 12-week intensity- and duration-graded aerobic training, three times in addition to the respiratory re-training. The G-AE program commenced with a training intensity corresponding to 50% of the maximum age-predicted heart rate for 25 minutes in the first two weeks, which progressed on a two-week basis, and ended up with a training intensity corresponding to 75% of the maximum age-predicted heart rate for 50 minutes in the last two weeks. The G-AE program also included a warm-up for 5 minutes and a cool-down for 5 minutes.
  Arms: G-AE group
Other: Respiratory Re-training — The respiratory re-training lasted for 30 minutes per session and was repeated three times a week for 12 consecutive weeks. The program consisted of diaphragmatic breathing exercises, breath-hold, and breathing control exercises, pursed lip breathing, respiratory muscle strengthening, postural correction exercises, and relaxation techniques.
  Arms: Control group

SUMMARY:
This study aimed to compare the effect of constant-load aerobic exercise (CL-AE) and graded aerobic exercise (G-AE) on cardiopulmonary fitness, and functional capacity in a cohort of obese children with bronchial asthma (BA).

A total of 78 children with BA were randomly assigned to the CL-AE group (n = 26, who underwent moderate-intensity aerobic training with the training load maintained at the same level throughout the entire program, besides the respiratory re-training program), the G-AE group (n = 26, received an intensity- and duration-graded aerobic training in addition to the respiratory re-training program), or the control group (n = 29, who only engaged in a respiratory re-training program). Interventions were administered three times/week for 12 successive weeks.

The cardiopulmonary fitness and functional capacity were evaluated in the three groups before and after the completion of the assigned interventions.

DETAILED DESCRIPTION:
Seventy-eight children with BA were recruited from the Pulmonary Medicine/Critical Care and Allergy-Immunology at King Khalid Hospital and two referral hospitals in Riyadh, Saudi Arabia. The study included children with moderate, clinically stable BA, aged 8-18 years, had a body mass index between 30 to 35 kg/m2, had no abnormalities of the lower limbs or spine, maintained constant medication dosages in the past three months, and did not engage in a regular exercise program (in the past six months). Children were excluded if they had exacerbated asthma symptoms, chronic lung comorbidities, and cardiovascular or musculoskeletal conditions expected to hinder the training.

Outcome measures

Cardiopulmonary fitness: The peak oxygen uptake was assessed through the McMaster cycling protocol.

Functional Capacity: The 6-minute walk test was used to assess the submaximal functional capacity Perceived dyspnea and fatigue: Borg's category ratio scale (CR-10) was used to explore how much dyspnea and fatigue they perceived after the 6-minute walk test.

Interventions

The CL-AE group received a 12-week aerobic training, three times in addition to the respiratory re-training. the program included a moderate-intensity aerobic training program, with an intensity set at 65% of the maximum age-predicted heart rate for 45 minutes. The training intensity and duration were maintained at the same level throughout the program. The CL-AE program included a warm-up for 5 minutes and a cool-down for 5 minutes.

The G-AE group received a 12-week aerobic training, three times in addition to the respiratory re-training. The G-AE program commenced with a training intensity corresponding to 50% of the maximum age-predicted heart rate for 25 minutes in the first two weeks, which progressed on a two-week basis, and ended up with a training intensity corresponding to 75% of the maximum age-predicted heart rate for 50 minutes in the last two weeks. The G-AE program also included a warm-up for 5 minutes and a cool-down for 5 minutes.

The control group received the respiratory re-training only, 30 minutes per session, three times a week for 12 consecutive weeks. The program consisted of diaphragmatic breathing exercises, breath-hold, and breathing control exercises, pursed lip breathing, respiratory muscle strengthening, postural correction exercises, and relaxation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age of 8-18 years
* Body mass index ranging from 30 to 35 kg/m2
* Verified asthma diagnosis per the Global Initiative for Asthma (GINA) criteria
* Moderate Onset
* Clinically Stable
* Maintained medication dosages in the past three months
* Free of lower limb or spinal deformities
* Not engaging in regular exercise regimens in the past six months.

Exclusion Criteria:

* Exacerbated asthma symptoms
* Chronic lung comorbidities
* Cardiovascular or musculoskeletal conditions expected to hinder the training.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | 3 months
  The peak oxygen uptake (mL/kg/min) was assessed through a symptom-free exercise tolerance test (i.e., the McMaster cycling protocol).

SECONDARY OUTCOMES:
Six-minute walk test | 3 months
  This test identified the maximum distance (m) that each child was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage.
Dyspnea | 3 months
  Dyspnea perception was assessed using Borg's category ratio scale (CR-10). Children rated the level of difficulty they experienced in breathing after completing the six-minute walk test on a 12-point scale. The scale ranges from 0 "no breathing difficulty" to 10 "maximal breathing difficulty".
Fatigue | 3 months
  Fatigue perception was evaluated using Borg's category ratio scale (CR-10). Children rated the level of exertion they felt after completing the six-minute walk test on a 12-point scale. The scale ranges from 0 "no fatigue" to 10 "significant fatigue".

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No